CLINICAL TRIAL: NCT01962805
Title: A Double-Blind, Crossover Study in Healthy Volunteers to Compare Two Formulations of Proellex for Vaginal Administration
Brief Title: Comparison of Two Formulations of Proellex for Vaginal Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ZPV-101
Record Dates: First submitted 2013-10-09; First posted 2013-10-14 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Comparison of 2 Different Formulations of 12 mg Proellex Vaginal Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proellex Schedule A (Experimental): Proellex vaginal capsule, 12 mg, once a day for up to 7 days
  Interventions: Drug: Proellex Formulation A; Drug: Proellex Formulation B
- Proellex Schedule B (Experimental): Proellex vaginal capsule, 12 mg, once a day for up to 7 days
  Interventions: Drug: Proellex Formulation A; Drug: Proellex Formulation B

INTERVENTIONS:
Drug: Proellex Formulation A
  Other Names: telepristone acetate
Drug: Proellex Formulation B
  Other Names: telepristone acetate

SUMMARY:
This study is a double-blind crossover study in female healthy volunteers to compare the pharmacokinetics and safety of either 1 or 6 days of dosing with two different formulations of Proellex for vaginal administration. Each formulation will be designated as either Treatment A or Treatment B. A total of 8 subjects who meet the eligibility criteria will be randomized to receive either Treatment A or Treatment B as their first assigned treatment. Subjects will receive a single dose of Treatment A or daily dosing with Treatment B for 6 days. After a 7-day washout period subjects will receive the alternative treatment. On the day of treatment with Treatment A and on the first and last days of treatment with Treatment B subjects will remain in the clinic overnight and undergo 32-hour pharmacokinetic assessment at the following time points: 0, 0.5, 1, 2, 4, 8, 12, 16, 20, 24, 28 and 32 hours after administration of study drug. For Treatment B study drug will be administered in the clinic each day after a trough blood sample has been drawn.

ELIGIBILITY:
Inclusion Criteria:

* Speak, read, and understand English or Spanish and is willing and able to provide written informed consent on an institutional review board (IRB)-approved form prior to the initiation of any study procedures;
* Healthy, premenopausal female age 18-47;
* History of menstrual events that occur in regular cycles
* Agreement not to attempt to become pregnant
* Agrees to use a condom and no other method of birth control (hormonal methods, contraceptive sponge, spermicide or cervical cap) over the course of the study;
* Has a negative pregnancy test at the Screening visit. An exception for the pregnancy test requirement will be granted for subjects reporting surgical sterilization in medical history
* Normal laboratory values or clinically insignificant findings at screening as determined by the Investigator;
* Subject is willing to remain in the clinic overnight for PK assessment on Days 0, 6 or 8 and Day 14.

Exclusion Criteria:

* Subject is a post-menopausal woman, defined as either; six (6) months or more (immediately prior to screening visit) without a menstrual period, or prior hysterectomy and/or oophorectomy
* Subject is pregnant or lactating or is attempting or expecting to become pregnant during the study
* Women with abnormally high liver enzymes or liver disease. Alanine transaminase (ALT) or aspartate aminotransferase (AST) exceeding 1.5 x upper limit of normal (ULN) AND total bilirubin exceeding 1.5 x ULN at screening and confirmed on repeat).
* Received an investigational drug in the 30 days prior to the screening for this study
* Women with a history of polycystic ovary syndrome (PCOS)
* Concurrent use of any testosterone, progestin, androgen, estrogen, anabolic steroids, dehydroepiandrosterone (DHEA) or hormonal products for at least 2 weeks prior to screening and during the study.
* Use of oral contraceptives in the preceding 2 weeks. Use of Depo-Provera® in the preceding 6 months.
* Has an intrauterine device (IUD) in place
* Women currently using narcotics
* Women currently taking spironolactone
* Infectious disease screen is positive for HIV or Hepatitis A, B or C.
* Clinically significant abnormal findings on screening examination or any condition which in the opinion of the investigator would interfere with the participant's ability to comply with the study instructions or endanger the participant if she took part in the study

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cmax | 7 days
  To determine and compare the maximum measured plasma concentration over the final dosing interval(Cmax) of two formulations of 12 mg Proellex administered vaginally in female healthy volunteers once daily for up to 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Houston, Texas, United States

REFERENCES:
- See also: Sponsor corporate website — http://www.reprosrx.com